CLINICAL TRIAL: NCT01038063
Title: Programmatic Implementation of ACTs in Malawi: Safety and Effectiveness of Combination Therapies With Repeated Treatments for Uncomplicated P. Falciparum Malaria Over a Three-year Period
Brief Title: Safety and Effectiveness of Artemisinin-based Combination Therapies (ACTs) With Repeated Treatments for Uncomplicated Falciparum Malaria Over a Three-year Period
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); National Malaria Control Programme, Malawi (Other Government); Research for Equity and Community Health Trust (Unknown)
Responsible Party: Sian Roberts / Head of Research Management, Liverpool School of Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.07
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Artemether-lumefantrine (Experimental): Children in this study arm will be treated with artemether-lumefantrine during a three year follow-up period each time a child develops uncomplicated malaria.
  Interventions: Drug: Artemether-lumefantrine combination
- Dihydroartemisinin-piperaquine (Active Comparator): Children in this study arm will be treated with dihydroartemisinin-piperaquine during a three year follow-up period each time a child develops uncomplicated malaria.
  Interventions: Drug: Artemether-lumefantrine combination

INTERVENTIONS:
Drug: Artemether-lumefantrine combination

SUMMARY:
A community-based, open-label, cluster-randomised longitudinal study in which children are randomized according to village health worker catchment areas comparing the safety and effectiveness of repeated treatments with artemether-lumefantrine (AL) over a 3-year period in children 4-48 months to that of repeated treatment with dihydroartemisinin-piperaquine (DHA-PPQ).

ELIGIBILITY:
Inclusion criteria

1. Aged between 4 months and 11 months at the time of randomization
2. Bodyweight ≥ 5 kg at the time of randomization
3. Provision of informed consent by parent or guardian
4. Intention to stay in the study area for the time of the study

Exclusion criteria

1. Ongoing participation into another clinical study involving ongoing or scheduled treatment with medicinal products
2. Intent to reside outside of catchment area during the course of the study
3. Known hypersensitivity to the study drug randomized to
4. Known pre-existing hearing problem or neurological impairment
5. Known need at the time of randomization for concomitant prohibited medication
6. Suspected non-compliance with the follow-up schedule

Ages: 4 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of ototoxicity at 18 months and 36 months of enrolment. | At 18 mo and 36 month of follow up

SECONDARY OUTCOMES:
Incidence of clinical malaria during 18 months and 36 months of follow-up | 18 and 36 months of follow up

CONTACTS AND LOCATIONS:
Overall Officials: David Lalloo, MD, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- Malawi-Liverpool-Wellcome Trust Research Programme, College of Medicine, Blantyre, Malawi

REFERENCES:
- [Derived] Roca-Feltrer A, Lalloo DG, Phiri K, Terlouw DJ. Rolling Malaria Indicator Surveys (rMIS): a potential district-level malaria monitoring and evaluation (M&E) tool for program managers. Am J Trop Med Hyg. 2012 Jan;86(1):96-8. doi: 10.4269/ajtmh.2012.11-0397. PMID 22232457